CLINICAL TRIAL: NCT00005176
Title: Long QT Syndrome-Population Genetics and Cardiac Studies
Acronym: LQTS
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arthur J. Moss, Professor, University of Rochester
Other Study IDs: 1053; R01HL033843-16 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Ventricular Arrhythmia; Long QT Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Long QT Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the clinical, genetic and cardiologic aspects of the Long QT Syndrome, a predominantly hereditary disease with episodic malignant arrhythmias and sudden death, and a demonstrated gene linkage in a large pedigree.

DETAILED DESCRIPTION:
BACKGROUND:

The Long QT Syndrome (LQTS) is an infrequently occurring disorder of unknown cause in which affected individuals have an unusual electrocardiographic repolarization abnormality and a propensity to syncope and fatal ventricular tachyarrhythmias. The first family with LQTS was described by Jervell and Lange-Nielsen in 1957. Three sudden deaths occurred in four deaf children with QT prolongation; two other children and the parents were healthy with normal hearing and normal electrocardiograms. The findings were interpreted as a pattern of autosomal recessive inheritance. Subsequent reports identified LQTS families with normal hearing (Romano-Ward Syndrome) having a pattern of occurrence suggesting autosomal dominant inheritance.

DESIGN NARRATIVE:

Beginning in 1985, patients and their unaffected relatives were longitudinally followed in this multicenter study to develop and validate widely applicable clinical criteria for stratifying the risk of life-threatening arrhythmias. A population of genetically deaf students was surveyed to identify additional families with the unique association of Long QT Syndrome and congenital deafness in order to expand the data base for genetic studies in the recessive form of the disorder, the Jervell and Lange-Nielsen Syndrome. Pedigrees of selected Long QT Syndrome families were recorded to better understand the inheritance of the dominant form of the disorder, the Romano-Ward Syndrome. Genetic studies were conducted using human leukocyte antigen and other protein markers in order to investigate the gene locus for the autosomal dominant form of the syndrome. A select group of 30 patients and 30 unaffected relatives had 24-hour Holter monitoring, treadmill exercise, Valsalva maneuver and handgrip stress tests to determine if the patients had a unique cardiovascular response to autonomic dysfunction.

The study was renewed in 1993. The renewal had six aims. The first examined genetic heterogeneity in LQTS by testing for Harvey-ras-1 gene linkage in the existing well-characterized LQTS families with evidence of a major gene by segregation analysis; in LQTS families that did not show Harvey-ras- 1 linkage, a search for other closely linked genetic markers was initiated. The second aim explored by segregation analysis the likelihood that a second gene coexisted with the Harvey-ras-1 gene to explain a more malignant disease process in some LQTS families than in others. The third established normal standards for six quantitative repolarization parameters on a healthy population (n=4,000) using digitized ECG recordings, and biomedical and statistical techniques with adjustment for age, gender, race, and heart rate. The fourth aim continued the existing LQTS registry with ongoing enrollment of new families and follow-up of new and existing LQTS pedigrees (n=370 families) in order to provide a central repository for this disorder, especially as it related to the natural history of this disorder and ongoing genetic analyses. The fifth aim investigated the static (12-lead ECG) and dynamic (24-hour Holter ECG) aspects of ventricular repolarization in LQTS families showing Harvey-ras gene linkage to upgrade the ECG categorization of delayed repolarization using the Harvey-ras- 1 marker as the gold standard to identify affected and unaffected individuals. The sixth aim continued the prospective longitudinal follow-up study of LQTS families to better understand the long-term clinical course of this disorder; time-dependent survivorship analyses were performed to evaluate the effects of various clinical features, repolarization severity (QTc length), Harvey-ras-I gene linkage, and therapeutic efficacy with antiadrenergic therapy (if data permits) on outcome event rates (syncope and sudden death) in the LQTS probands.

The study has been renewed several times to: expand the pedigrees of LQTS families and family members enrolled in the registry; identify new LQTS gene mutations and expand the number of gene-identified affected and unaffected members in LQTS families with known gene mutations; investigate phenotype-genotype relationships in 200 genotyped families involving 1,200 affected and unaffected family members regarding the clinical course of LQTS, T-wave repolarization, triggering factors for cardiac events, and co-morbidity associations, all by genotype. The study remains a multicenter project with six clinical centers, a genetic component involving four molecular genetic labs, a statistical genetic component, a biostatistical component, and a coordinating center.

ELIGIBILITY:
Probands are required to have clinical dx of LQTS. Family members are also invited to participate regardless of their dx.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As of the 2013 closeout report, 1329 probands with clinical dx of LQTS and members of their extended families have been enrolled in the LQTS Registry. By ECG classification, this includes 3420 probands and affected family members, 3533 unaffected family members, and 2105 family members with borderline QTc. Of those, 2125 have had mutations identified.
Sampling Method: Non-Probability Sample
Enrollment: 2125 (Actual)
Dates: Start 1985-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
None. This is an observational study. | By study end

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Moss, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Weitkamp LR, Moss AJ: The Long QT (Romano-Ward) Syndrome Locus, LQT, is Probably Linked to the HLA Loci. Cytogenet Cell Genet, 40:775, 1985
- [Background] Locati E, Schwartz PJ, Moss AJ, Crampton RS: Long-Term Survival After Left Cervico-Thoracic Sympathectomy in High Risk Long QT Syndrome Patients With Refractory Ventricular Arrhythmias. J Am Coll Cardiol, 7:234A, 1986
- [Background] De Ambroggi L, Bertoni T, Locati E, Stramba-Badiale M, Schwartz PJ. Mapping of body surface potentials in patients with the idiopathic long QT syndrome. Circulation. 1986 Dec;74(6):1334-45. doi: 10.1161/01.cir.74.6.1334. PMID 3779919
- [Background] Vincent GM. The heart rate of Romano-Ward syndrome patients. Am Heart J. 1986 Jul;112(1):61-4. doi: 10.1016/0002-8703(86)90678-2. PMID 3728288
- [Background] Moss AJ. Prolonged QT-interval syndromes. JAMA. 1986 Dec 5;256(21):2985-7. No abstract available. PMID 3773216
- [Background] Merri M, Benhorin J, Alberti M, Locati E, Moss AJ. Electrocardiographic quantitation of ventricular repolarization. Circulation. 1989 Nov;80(5):1301-8. doi: 10.1161/01.cir.80.5.1301. PMID 2805266
- [Background] Benhorin J, Merri M, Alberti M, Locati E, Moss AJ, Hall WJ, Cui L. Long QT syndrome. New electrocardiographic characteristics. Circulation. 1990 Aug;82(2):521-7. doi: 10.1161/01.cir.82.2.521. PMID 2271025
- [Background] Moss AJ. Clinical management of patients with the long QT syndrome: drugs, devices, and gene-specific therapy. Pacing Clin Electrophysiol. 1997 Aug;20(8 Pt 2):2058-60. doi: 10.1111/j.1540-8159.1997.tb03627.x. PMID 9272508
- [Background] Zareba W, Moss AJ, le Cessie S, Locati EH, Robinson JL, Hall WJ, Andrews ML. Risk of cardiac events in family members of patients with long QT syndrome. J Am Coll Cardiol. 1995 Dec;26(7):1685-91. doi: 10.1016/0735-1097(95)60383-2. PMID 7594104
- [Background] Weitkamp LR, Moss AJ, Lewis RA, Hall WJ, MacCluer JW, Schwartz PJ, Locati EH, Tzivoni D, Vincent GM, Robinson JL, et al. Analysis of HLA and disease susceptibility: chromosome 6 genes and sex influence long-QT phenotype. Am J Hum Genet. 1994 Dec;55(6):1230-41. PMID 7977384
- [Background] Malfatto G, Beria G, Sala S, Bonazzi O, Schwartz PJ. Quantitative analysis of T wave abnormalities and their prognostic implications in the idiopathic long QT syndrome. J Am Coll Cardiol. 1994 Feb;23(2):296-301. doi: 10.1016/0735-1097(94)90410-3. PMID 7905012
- [Background] Zareba W, Moss AJ, le Cessie S, Hall WJ. T wave alternans in idiopathic long QT syndrome. J Am Coll Cardiol. 1994 Jun;23(7):1541-6. doi: 10.1016/0735-1097(94)90653-x. PMID 8195511
- [Background] Schwartz PJ, Priori SG, Locati EH, Napolitano C, Cantu F, Towbin JA, Keating MT, Hammoude H, Brown AM, Chen LS, Colatsky TJ. Long QT syndrome patients with mutations of the SCN5A and HERG genes have differential responses to Na+ channel blockade and to increases in heart rate. Implications for gene-specific therapy. Circulation. 1995 Dec 15;92(12):3381-6. doi: 10.1161/01.cir.92.12.3381. PMID 8521555
- [Background] De Ferrari GM, Nador F, Beria G, Sala S, Lotto A, Schwartz PJ. Effect of calcium channel block on the wall motion abnormality of the idiopathic long QT syndrome. Circulation. 1994 May;89(5):2126-32. doi: 10.1161/01.cir.89.5.2126. PMID 8181137
- [Background] Wang Q, Shen J, Splawski I, Atkinson D, Li Z, Robinson JL, Moss AJ, Towbin JA, Keating MT. SCN5A mutations associated with an inherited cardiac arrhythmia, long QT syndrome. Cell. 1995 Mar 10;80(5):805-11. doi: 10.1016/0092-8674(95)90359-3. PMID 7889574
- [Background] Moss AJ. Measurement of the QT interval and the risk associated with QTc interval prolongation: a review. Am J Cardiol. 1993 Aug 26;72(6):23B-25B. doi: 10.1016/0002-9149(93)90036-c. PMID 8256751
- [Background] Schwartz PJ, Moss AJ, Vincent GM, Crampton RS. Diagnostic criteria for the long QT syndrome. An update. Circulation. 1993 Aug;88(2):782-4. doi: 10.1161/01.cir.88.2.782. No abstract available. PMID 8339437
- [Background] Moss AJ, Robinson JL. Clinical aspects of the idiopathic long QT syndrome. Ann N Y Acad Sci. 1992 Jan 27;644:103-11. doi: 10.1111/j.1749-6632.1992.tb31006.x. No abstract available. PMID 1348608
- [Background] Moss AJ, Robinson J. Clinical features of the idiopathic long QT syndrome. Circulation. 1992 Jan;85(1 Suppl):I140-4. PMID 1345816
- [Background] Merri M, Moss AJ, Benhorin J, Locati EH, Alberti M, Badilini F. Relation between ventricular repolarization duration and cardiac cycle length during 24-hour Holter recordings. Findings in normal patients and patients with long QT syndrome. Circulation. 1992 May;85(5):1816-21. doi: 10.1161/01.cir.85.5.1816. PMID 1572038
- [Background] Nador F, Beria G, De Ferrari GM, Stramba-Badiale M, Locati EH, Lotto A, Schwartz PJ. Unsuspected echocardiographic abnormality in the long QT syndrome. Diagnostic, prognostic, and pathogenetic implications. Circulation. 1991 Oct;84(4):1530-42. doi: 10.1161/01.cir.84.4.1530. PMID 1914095
- [Background] Moss AJ, Liu JE, Gottlieb S, Locati EH, Schwartz PJ, Robinson JL. Efficacy of permanent pacing in the management of high-risk patients with long QT syndrome. Circulation. 1991 Oct;84(4):1524-9. doi: 10.1161/01.cir.84.4.1524. PMID 1914094
- [Background] Moss AJ, Schwartz PJ, Crampton RS, Tzivoni D, Locati EH, MacCluer J, Hall WJ, Weitkamp L, Vincent GM, Garson A Jr, et al. The long QT syndrome. Prospective longitudinal study of 328 families. Circulation. 1991 Sep;84(3):1136-44. doi: 10.1161/01.cir.84.3.1136. PMID 1884444
- [Background] De Ambroggi L, Negroni MS, Monza E, Bertoni T, Schwartz PJ. Dispersion of ventricular repolarization in the long QT syndrome. Am J Cardiol. 1991 Sep 1;68(6):614-20. doi: 10.1016/0002-9149(91)90353-m. PMID 1877478
- [Background] Schwartz PJ, Locati EH, Moss AJ, Crampton RS, Trazzi R, Ruberti U. Left cardiac sympathetic denervation in the therapy of congenital long QT syndrome. A worldwide report. Circulation. 1991 Aug;84(2):503-11. doi: 10.1161/01.cir.84.2.503. PMID 1860195
- [Background] Schwartz PJ, Zaza A, Locati E, Moss AJ. Stress and sudden death. The case of the long QT syndrome. Circulation. 1991 Apr;83(4 Suppl):II71-80. PMID 2009631
- [Background] Moss AJ, Merri M, Benhorin J, Alberti M, Locati E. Multidimensional quantitation of ventricular repolarization. Static and dynamic characteristics. Ann N Y Acad Sci. 1990;601:31-5. doi: 10.1111/j.1749-6632.1990.tb37289.x. No abstract available. PMID 2221694
- [Background] Curran M, Atkinson D, Timothy K, Vincent GM, Moss AJ, Leppert M, Keating M. Locus heterogeneity of autosomal dominant long QT syndrome. J Clin Invest. 1993 Aug;92(2):799-803. doi: 10.1172/JCI116653. PMID 8102381
- [Background] Rashba EJ, Zareba W, Moss AJ, Hall WJ, Robinson J, Locati EH, Schwartz PJ, Andrews M. Influence of pregnancy on the risk for cardiac events in patients with hereditary long QT syndrome. LQTS Investigators. Circulation. 1998 Feb 10;97(5):451-6. doi: 10.1161/01.cir.97.5.451. PMID 9490239
- [Background] Locati EH, Zareba W, Moss AJ, Schwartz PJ, Vincent GM, Lehmann MH, Towbin JA, Priori SG, Napolitano C, Robinson JL, Andrews M, Timothy K, Hall WJ. Age- and sex-related differences in clinical manifestations in patients with congenital long-QT syndrome: findings from the International LQTS Registry. Circulation. 1998 Jun 9;97(22):2237-44. doi: 10.1161/01.cir.97.22.2237. PMID 9631873
- [Background] Benhorin J, Taub R, Goldmit M, Kerem B, Kass RS, Windman I, Medina A. Effects of flecainide in patients with new SCN5A mutation: mutation-specific therapy for long-QT syndrome? Circulation. 2000 Apr 11;101(14):1698-706. doi: 10.1161/01.cir.101.14.1698. PMID 10758053
- [Background] Ali RH, Zareba W, Moss AJ, Schwartz PJ, Benhorin J, Vincent GM, Locati EH, Priori S, Napolitano C, Towbin JA, Hall WJ, Robinson JL, Andrews ML, Zhang L, Timothy K, Medina A. Clinical and genetic variables associated with acute arousal and nonarousal-related cardiac events among subjects with long QT syndrome. Am J Cardiol. 2000 Feb 15;85(4):457-61. doi: 10.1016/s0002-9149(99)90772-5. PMID 10728950
- [Background] Moss AJ, Zareba W, Hall WJ, Schwartz PJ, Crampton RS, Benhorin J, Vincent GM, Locati EH, Priori SG, Napolitano C, Medina A, Zhang L, Robinson JL, Timothy K, Towbin JA, Andrews ML. Effectiveness and limitations of beta-blocker therapy in congenital long-QT syndrome. Circulation. 2000 Feb 15;101(6):616-23. doi: 10.1161/01.cir.101.6.616. PMID 10673253
- [Background] Benhorin J, Goldmit M, MacCluer JW, Blangero J, Goffen R, Leibovitch A, Rahat A, Wang Q, Medina A, Towbin J, Kerem B. Identification of a new SCN5A mutation, D1840G, associated with the long QT syndrome. Mutations in brief no. 153. Online. Hum Mutat. 1998;12(1):72. doi: 10.1002/(SICI)1098-1004(1998)12:13.0.CO;2-T. PMID 10627139
- [Background] Rosero SZ, Zareba W, Moss AJ, Robinson JL, Hajj Ali RH, Locati EH, Benhorin J, Andrews ML. Asthma and the risk of cardiac events in the Long QT syndrome. Long QT Syndrome Investigative Group. Am J Cardiol. 1999 Dec 15;84(12):1406-11. doi: 10.1016/s0002-9149(99)00586-x. PMID 10606113
- [Background] Couderc JP, Zareba W, Burattini L, Moss AJ. Beat-to-Beat repolarization variability in LQTS patients with the SCN5A sodium channel gene mutation. Pacing Clin Electrophysiol. 1999 Nov;22(11):1581-92. doi: 10.1111/j.1540-8159.1999.tb00376.x. PMID 10598960
- [Background] Moss AJ, Robinson JL, Gessman L, Gillespie R, Zareba W, Schwartz PJ, Vincent GM, Benhorin J, Heilbron EL, Towbin JA, Priori SG, Napolitano C, Zhang L, Medina A, Andrews ML, Timothy K. Comparison of clinical and genetic variables of cardiac events associated with loud noise versus swimming among subjects with the long QT syndrome. Am J Cardiol. 1999 Oct 15;84(8):876-9. doi: 10.1016/s0002-9149(99)00458-0. PMID 10532503
- [Background] Chen Q, Zhang D, Gingell RL, Moss AJ, Napolitano C, Priori SG, Schwartz PJ, Kehoe E, Robinson JL, Schulze-Bahr E, Wang Q, Towbin JA. Homozygous deletion in KVLQT1 associated with Jervell and Lange-Nielsen syndrome. Circulation. 1999 Mar 16;99(10):1344-7. doi: 10.1161/01.cir.99.10.1344. PMID 10077519
- [Background] Couderc JP, Zareba W, Burattini L, Konecki JA, Moss AJ. Beat-to-beat repolarization variability in amplitude and duration in LQTS patients with the SCN5A sodium channel gene mutation. J Electrocardiol. 1998;31 Suppl:134. doi: 10.1016/s0022-0736(98)90306-5. No abstract available. PMID 9988018
- [Background] Zareba W, Moss AJ, Schwartz PJ, Vincent GM, Robinson JL, Priori SG, Benhorin J, Locati EH, Towbin JA, Keating MT, Lehmann MH, Hall WJ. Influence of the genotype on the clinical course of the long-QT syndrome. International Long-QT Syndrome Registry Research Group. N Engl J Med. 1998 Oct 1;339(14):960-5. doi: 10.1056/NEJM199810013391404. PMID 9753711
- [Background] Moss AJ. Management of patients with the hereditary long QT syndrome. J Cardiovasc Electrophysiol. 1998 Jun;9(6):668-74. doi: 10.1111/j.1540-8167.1998.tb00952.x. PMID 9654236
- [Background] Li H, Chen Q, Moss AJ, Robinson J, Goytia V, Perry JC, Vincent GM, Priori SG, Lehmann MH, Denfield SW, Duff D, Kaine S, Shimizu W, Schwartz PJ, Wang Q, Towbin JA. New mutations in the KVLQT1 potassium channel that cause long-QT syndrome. Circulation. 1998 Apr 7;97(13):1264-9. doi: 10.1161/01.cir.97.13.1264. PMID 9570196
- [Background] Moss AJ. The long QT syndrome revisited: current understanding and implications for treatment. Pacing Clin Electrophysiol. 1997 Dec;20(12 Pt 1):2879-81. doi: 10.1111/j.1540-8159.1997.tb05455.x. No abstract available. PMID 9455746
- [Background] Schwartz PJ, Priori SG, Spazzolini C, Moss AJ, Vincent GM, Napolitano C, Denjoy I, Guicheney P, Breithardt G, Keating MT, Towbin JA, Beggs AH, Brink P, Wilde AA, Toivonen L, Zareba W, Robinson JL, Timothy KW, Corfield V, Wattanasirichaigoon D, Corbett C, Haverkamp W, Schulze-Bahr E, Lehmann MH, Schwartz K, Coumel P, Bloise R. Genotype-phenotype correlation in the long-QT syndrome: gene-specific triggers for life-threatening arrhythmias. Circulation. 2001 Jan 2;103(1):89-95. doi: 10.1161/01.cir.103.1.89. PMID 11136691
- [Background] Splawski I, Shen J, Timothy KW, Lehmann MH, Priori S, Robinson JL, Moss AJ, Schwartz PJ, Towbin JA, Vincent GM, Keating MT. Spectrum of mutations in long-QT syndrome genes. KVLQT1, HERG, SCN5A, KCNE1, and KCNE2. Circulation. 2000 Sep 5;102(10):1178-85. doi: 10.1161/01.cir.102.10.1178. PMID 10973849
- [Background] Jiang C, Atkinson D, Towbin JA, Splawski I, Lehmann MH, Li H, Timothy K, Taggart RT, Schwartz PJ, Vincent GM, et al. Two long QT syndrome loci map to chromosomes 3 and 7 with evidence for further heterogeneity. Nat Genet. 1994 Oct;8(2):141-7. doi: 10.1038/ng1094-141. PMID 7842012
- [Background] Benhorin J, Moss AJ, Bak M, Zareba W, Kaufman ES, Kerem B, Towbin JA, Priori S, Kass RS, Attali B, Brown AM, Ficker E. Variable expression of long QT syndrome among gene carriers from families with five different HERG mutations. Ann Noninvasive Electrocardiol. 2002 Jan;7(1):40-6. doi: 10.1111/j.1542-474x.2001.tb00137.x. PMID 11844290
- [Background] Perkiomaki JS, Zareba W, Couderc JP, Moss AJ. Heart rate variability in patients with congenital long QT syndrome. Ann Noninvasive Electrocardiol. 2001 Oct;6(4):298-304. doi: 10.1111/j.1542-474x.2001.tb00122.x. PMID 11686910
- [Background] Kimbrough J, Moss AJ, Zareba W, Robinson JL, Hall WJ, Benhorin J, Locati EH, Medina A, Napolitano C, Priori S, Schwartz PJ, Timothy K, Towbin JA, Vincent GM, Zhang L. Clinical implications for affected parents and siblings of probands with long-QT syndrome. Circulation. 2001 Jul 31;104(5):557-62. doi: 10.1161/hc3001.093501. PMID 11479253
- [Background] Windle JR, Geletka RC, Moss AJ, Zareba W, Atkins DL. Normalization of ventricular repolarization with flecainide in long QT syndrome patients with SCN5A:DeltaKPQ mutation. Ann Noninvasive Electrocardiol. 2001 Apr;6(2):153-8. doi: 10.1111/j.1542-474x.2001.tb00100.x. PMID 11333173
- [Background] Wang Z, Li H, Moss AJ, Robinson J, Zareba W, Knilans T, Bowles NE, Towbin JA. Compound heterozygous mutations in KvLQT1 cause Jervell and Lange-Nielsen syndrome. Mol Genet Metab. 2002 Apr;75(4):308-16. doi: 10.1016/S1096-7192(02)00007-0. PMID 12051962
- [Background] Perkiomaki JS, Zareba W, Nomura A, Andrews M, Kaufman ES, Moss AJ. Repolarization dynamics in patients with long QT syndrome. J Cardiovasc Electrophysiol. 2002 Jul;13(7):651-6. doi: 10.1046/j.1540-8167.2002.00651.x. PMID 12139286
- [Background] Moss AJ. Long QT Syndrome. JAMA. 2003 Apr 23-30;289(16):2041-4. doi: 10.1001/jama.289.16.2041. No abstract available. PMID 12709446
- [Background] Moss AJ. T-wave patterns associated with the hereditary long QT syndrome. Card Electrophysiol Rev. 2002 Sep;6(3):311-5. doi: 10.1023/a:1016301730302. PMID 12114857
- [Background] Kupershmidt S, Yang T, Chanthaphaychith S, Wang Z, Towbin JA, Roden DM. Defective human Ether-a-go-go-related gene trafficking linked to an endoplasmic reticulum retention signal in the C terminus. J Biol Chem. 2002 Jul 26;277(30):27442-8. doi: 10.1074/jbc.M112375200. Epub 2002 May 20. PMID 12021266
- [Background] Zareba W, Moss AJ, Sheu G, Kaufman ES, Priori S, Vincent GM, Towbin JA, Benhorin J, Schwartz PJ, Napolitano C, Hall WJ, Keating MT, Qi M, Robinson J, Andrews ML; International LQTS Registry, University of Rochester, Rochester, New York. Location of mutation in the KCNQ1 and phenotypic presentation of long QT syndrome. J Cardiovasc Electrophysiol. 2003 Nov;14(11):1149-53. doi: 10.1046/j.1540-8167.2003.03177.x. PMID 14678125
- [Background] Ning L, Moss A, Zareba W, Robinson J, Rosero S, Ryan D, Qi M. Denaturing high-performance liquid chromatography quickly and reliably detects cardiac ion channel mutations in long QT syndrome. Genet Test. 2003 Fall;7(3):249-53. doi: 10.1089/109065703322537287. PMID 14642002
- [Background] Ning L, Moss AJ, Zareba W, Robinson J, Rosero S, Ryan D, Qi M. Novel compound heterozygous mutations in the KCNQ1 gene associated with autosomal recessive long QT syndrome (Jervell and Lange-Nielsen syndrome). Ann Noninvasive Electrocardiol. 2003 Jul;8(3):246-50. doi: 10.1046/j.1542-474x.2003.08313.x. PMID 14510661
- [Background] Zareba W, Moss AJ, Locati EH, Lehmann MH, Peterson DR, Hall WJ, Schwartz PJ, Vincent GM, Priori SG, Benhorin J, Towbin JA, Robinson JL, Andrews ML, Napolitano C, Timothy K, Zhang L, Medina A; International Long QT Syndrome Registry. Modulating effects of age and gender on the clinical course of long QT syndrome by genotype. J Am Coll Cardiol. 2003 Jul 2;42(1):103-9. doi: 10.1016/s0735-1097(03)00554-0. PMID 12849668
- [Background] Schwartz PJ, Priori SG, Cerrone M, Spazzolini C, Odero A, Napolitano C, Bloise R, De Ferrari GM, Klersy C, Moss AJ, Zareba W, Robinson JL, Hall WJ, Brink PA, Toivonen L, Epstein AE, Li C, Hu D. Left cardiac sympathetic denervation in the management of high-risk patients affected by the long-QT syndrome. Circulation. 2004 Apr 20;109(15):1826-33. doi: 10.1161/01.CIR.0000125523.14403.1E. Epub 2004 Mar 29. PMID 15051644
- [Background] Moss AJ, Schwartz PJ. 25th anniversary of the International Long-QT Syndrome Registry: an ongoing quest to uncover the secrets of long-QT syndrome. Circulation. 2005 Mar 8;111(9):1199-201. doi: 10.1161/01.CIR.0000157069.91834.DA. No abstract available. PMID 15753228
- [Background] Goldenberg I, Bradley J, Moss A, McNitt S, Polonsky S, Robinson JL, Andrews M, Zareba W; International LQTS Registry Investigators. Beta-blocker efficacy in high-risk patients with the congenital long-QT syndrome types 1 and 2: implications for patient management. J Cardiovasc Electrophysiol. 2010 Aug 1;21(8):893-901. doi: 10.1111/j.1540-8167.2010.01737.x. Epub 2010 Mar 5. PMID 20233272
- [Background] Horr S, Goldenberg I, Moss AJ, O-Uchi J, Barsheshet A, Connelly H, Gray DA, Zareba W, Lopes CM. Ion channel mechanisms related to sudden cardiac death in phenotype-negative long-QT syndrome genotype-phenotype correlations of the KCNQ1(S349W) mutation. J Cardiovasc Electrophysiol. 2011 Feb;22(2):193-200. doi: 10.1111/j.1540-8167.2010.01852.x. PMID 20662986
- [Background] Moss AJ. Sex hormones and ventricular tachyarrhythmias in LQTS: new insights regarding antiarrhythmic therapy. Heart Rhythm. 2012 May;9(5):833-4. doi: 10.1016/j.hrthm.2012.01.014. Epub 2012 Jan 20. No abstract available. PMID 22266129
- [Background] Goldenberg I, Thottathil P, Lopes CM, Moss AJ, McNitt S, O-Uchi J, Robinson JL, Zareba W, Ackerman MJ, Kaufman ES, Towbin JA, Vincent M, Barsheshet A. Trigger-specific ion-channel mechanisms, risk factors, and response to therapy in type 1 long QT syndrome. Heart Rhythm. 2012 Jan;9(1):49-56. doi: 10.1016/j.hrthm.2011.08.020. Epub 2011 Aug 24. PMID 21871251
- [Background] Barsheshet A, Moss AJ, McNitt S, Polonsky S, Lopes CM, Zareba W, Robinson JL, Ackerman MJ, Benhorin J, Kaufman ES, Towbin JA, Vincent GM, Qi M, Goldenberg I. Risk of syncope in family members who are genotype-negative for a family-associated long-QT syndrome mutation. Circ Cardiovasc Genet. 2011 Oct;4(5):491-9. doi: 10.1161/CIRCGENETICS.111.960179. Epub 2011 Aug 10. PMID 21831960
- [Background] Migdalovich D, Moss AJ, Lopes CM, Costa J, Ouellet G, Barsheshet A, McNitt S, Polonsky S, Robinson JL, Zareba W, Ackerman MJ, Benhorin J, Kaufman ES, Platonov PG, Shimizu W, Towbin JA, Vincent GM, Wilde AA, Goldenberg I. Mutation and gender-specific risk in type 2 long QT syndrome: implications for risk stratification for life-threatening cardiac events in patients with long QT syndrome. Heart Rhythm. 2011 Oct;8(10):1537-43. doi: 10.1016/j.hrthm.2011.03.049. Epub 2011 Mar 25. PMID 21440677
- [Background] Barsheshet A, Peterson DR, Moss AJ, Schwartz PJ, Kaufman ES, McNitt S, Polonsky S, Buber J, Zareba W, Robinson JL, Ackerman MJ, Benhorin J, Towbin JA, Vincent GM, Zhang L, Goldenberg I. Genotype-specific QT correction for heart rate and the risk of life-threatening cardiac events in adolescents with congenital long-QT syndrome. Heart Rhythm. 2011 Aug;8(8):1207-13. doi: 10.1016/j.hrthm.2011.03.009. Epub 2011 Mar 10. PMID 21397043
- [Background] Couderc JP, Xia X, Peterson DR, McNitt S, Zhao H, Polonsky S, Moss AJ, Zareba W. T-wave morphology abnormalities in benign, potent, and arrhythmogenic I(kr) inhibition. Heart Rhythm. 2011 Jul;8(7):1036-43. doi: 10.1016/j.hrthm.2011.02.005. Epub 2011 Feb 9. PMID 21315844
- [Background] Patrick CC, Goust JM, Virella G. Tolerance and autoimmunity. Immunol Ser. 1990;50:415-33. No abstract available. PMID 2151124
- [Background] Liu JF, Jons C, Moss AJ, McNitt S, Peterson DR, Qi M, Zareba W, Robinson JL, Barsheshet A, Ackerman MJ, Benhorin J, Kaufman ES, Locati EH, Napolitano C, Priori SG, Schwartz PJ, Towbin J, Vincent M, Zhang L, Goldenberg I; International Long QT Syndrome Registry. Risk factors for recurrent syncope and subsequent fatal or near-fatal events in children and adolescents with long QT syndrome. J Am Coll Cardiol. 2011 Feb 22;57(8):941-50. doi: 10.1016/j.jacc.2010.10.025. PMID 21329841
- [Background] Goldenberg I, Horr S, Moss AJ, Lopes CM, Barsheshet A, McNitt S, Zareba W, Andrews ML, Robinson JL, Locati EH, Ackerman MJ, Benhorin J, Kaufman ES, Napolitano C, Platonov PG, Priori SG, Qi M, Schwartz PJ, Shimizu W, Towbin JA, Vincent GM, Wilde AA, Zhang L. Risk for life-threatening cardiac events in patients with genotype-confirmed long-QT syndrome and normal-range corrected QT intervals. J Am Coll Cardiol. 2011 Jan 4;57(1):51-9. doi: 10.1016/j.jacc.2010.07.038. PMID 21185501
- [Background] Zareba W. Counting mRNA in blood of LQTS - new direction? Kardiol Pol. 2011;69(5):430. No abstract available. PMID 21594823
- [Background] Kim JA, Lopes CM, Moss AJ, McNitt S, Barsheshet A, Robinson JL, Zareba W, Ackerman MJ, Kaufman ES, Towbin JA, Vincent M, Goldenberg I. Trigger-specific risk factors and response to therapy in long QT syndrome type 2. Heart Rhythm. 2010 Dec;7(12):1797-805. doi: 10.1016/j.hrthm.2010.09.011. Epub 2010 Sep 17. PMID 20850565
- [Background] Zhang T, Moss A, Cong P, Pan M, Chang B, Zheng L, Fang Q, Zareba W, Robinson J, Lin C, Li Z, Wei J, Zeng Q; Long QT International Registry Investigators; HVP-China Investigators; Qi M. LQTS gene LOVD database. Hum Mutat. 2010 Nov;31(11):E1801-10. doi: 10.1002/humu.21341. PMID 20809527
- [Background] Jons C, Moss AJ, Goldenberg I, Liu J, McNitt S, Zareba W, Qi M, Robinson JL. Risk of fatal arrhythmic events in long QT syndrome patients after syncope. J Am Coll Cardiol. 2010 Feb 23;55(8):783-8. doi: 10.1016/j.jacc.2009.11.042. PMID 20170817
- [Background] Ouellet G, Moss AJ, Jons C, McNitt S, Mullally J, Fugate T, Goldenberg I, Zareba W, Robinson JL; Investigators from the U.S. Portion of the International Long QT Syndrome Registry. Influence of diabetes mellitus on outcome in patients over 40 years of age with the long QT syndrome. Am J Cardiol. 2010 Jan 1;105(1):87-9. doi: 10.1016/j.amjcard.2009.08.657. Epub 2009 Oct 23. PMID 20102896
- [Background] Fugate T 2nd, Moss AJ, Jons C, McNitt S, Mullally J, Ouellet G, Goldenberg I, Zareba W, Robinson JL; U.S. portion of International Long QT Syndrome Registry Investigators. Long QT syndrome in African-Americans. Ann Noninvasive Electrocardiol. 2010 Jan;15(1):73-6. doi: 10.1111/j.1542-474X.2009.00342.x. PMID 20146785
- [Background] Shimizu W, Moss AJ, Wilde AA, Towbin JA, Ackerman MJ, January CT, Tester DJ, Zareba W, Robinson JL, Qi M, Vincent GM, Kaufman ES, Hofman N, Noda T, Kamakura S, Miyamoto Y, Shah S, Amin V, Goldenberg I, Andrews ML, McNitt S. Genotype-phenotype aspects of type 2 long QT syndrome. J Am Coll Cardiol. 2009 Nov 24;54(22):2052-62. doi: 10.1016/j.jacc.2009.08.028. PMID 19926013
- [Background] Spazzolini C, Mullally J, Moss AJ, Schwartz PJ, McNitt S, Ouellet G, Fugate T, Goldenberg I, Jons C, Zareba W, Robinson JL, Ackerman MJ, Benhorin J, Crotti L, Kaufman ES, Locati EH, Qi M, Napolitano C, Priori SG, Towbin JA, Vincent GM. Clinical implications for patients with long QT syndrome who experience a cardiac event during infancy. J Am Coll Cardiol. 2009 Aug 25;54(9):832-7. doi: 10.1016/j.jacc.2009.05.029. PMID 19695463
- [Background] Lane RD, Reis HT, Peterson DR, Zareba W, Moss AJ. Happiness and stress alter susceptibility to cardiac events in Long QT Syndrome. Ann Noninvasive Electrocardiol. 2009 Apr;14(2):193-200. doi: 10.1111/j.1542-474X.2009.00295.x. PMID 19419405
- [Background] Goldenberg I, Zareba W, Moss AJ. Long QT Syndrome. Curr Probl Cardiol. 2008 Nov;33(11):629-94. doi: 10.1016/j.cpcardiol.2008.07.002. PMID 18835466
- [Background] Zareba W, Cygankiewicz I. Long QT syndrome and short QT syndrome. Prog Cardiovasc Dis. 2008 Nov-Dec;51(3):264-78. doi: 10.1016/j.pcad.2008.10.006. PMID 19026859
- [Background] Thottathil P, Acharya J, Moss AJ, Jons C, McNitt S, Goldenberg I, Zareba W, Kaufman E, Qi M, Robinson JL; International Long QT Syndrome Investigative Group. Risk of cardiac events in patients with asthma and long-QT syndrome treated with beta(2) agonists. Am J Cardiol. 2008 Oct 1;102(7):871-4. doi: 10.1016/j.amjcard.2008.05.029. Epub 2008 Jul 17. PMID 18805113
- [Background] Sze E, Moss AJ, Goldenberg I, McNitt S, Jons C, Zareba W, Qi M, Robinson JL; International Long QT Syndrome Investigative Group. Long QT syndrome in patients over 40 years of age: increased risk for LQTS-related cardiac events in patients with coronary disease. Ann Noninvasive Electrocardiol. 2008 Oct;13(4):327-31. doi: 10.1111/j.1542-474X.2008.00250.x. PMID 18973489
- [Background] Wu G, Ai T, Kim JJ, Mohapatra B, Xi Y, Li Z, Abbasi S, Purevjav E, Samani K, Ackerman MJ, Qi M, Moss AJ, Shimizu W, Towbin JA, Cheng J, Vatta M. alpha-1-syntrophin mutation and the long-QT syndrome: a disease of sodium channel disruption. Circ Arrhythm Electrophysiol. 2008 Aug;1(3):193-201. doi: 10.1161/CIRCEP.108.769224. PMID 19684871
- [Background] Liu JF, Goldenberg I, Moss AJ, Shimizu W, Wilde AA, Hofman N, McNitt S, Zareba W, Miyamato Y, Robinson JL, Andrews ML. Phenotypic variability in Caucasian and Japanese patients with matched LQT1 mutations. Ann Noninvasive Electrocardiol. 2008 Jul;13(3):234-41. doi: 10.1111/j.1542-474X.2008.00226.x. PMID 18713323
- [Background] Goldenberg I, Moss AJ. Long QT syndrome. J Am Coll Cardiol. 2008 Jun 17;51(24):2291-300. doi: 10.1016/j.jacc.2008.02.068. PMID 18549912
- [Background] Kaufman ES, McNitt S, Moss AJ, Zareba W, Robinson JL, Hall WJ, Ackerman MJ, Benhorin J, Locati ET, Napolitano C, Priori SG, Schwartz PJ, Towbin JA, Vincent GM, Zhang L. Risk of death in the long QT syndrome when a sibling has died. Heart Rhythm. 2008 Jun;5(6):831-6. doi: 10.1016/j.hrthm.2008.02.029. Epub 2008 Mar 4. PMID 18534367
- [Background] Goldenberg I, Moss AJ, Peterson DR, McNitt S, Zareba W, Andrews ML, Robinson JL, Locati EH, Ackerman MJ, Benhorin J, Kaufman ES, Napolitano C, Priori SG, Qi M, Schwartz PJ, Towbin JA, Vincent GM, Zhang L. Risk factors for aborted cardiac arrest and sudden cardiac death in children with the congenital long-QT syndrome. Circulation. 2008 Apr 29;117(17):2184-91. doi: 10.1161/CIRCULATIONAHA.107.701243. Epub 2008 Apr 21. PMID 18427136
- [Background] Goldenberg I, Moss AJ, Bradley J, Polonsky S, Peterson DR, McNitt S, Zareba W, Andrews ML, Robinson JL, Ackerman MJ, Benhorin J, Kaufman ES, Locati EH, Napolitano C, Priori SG, Qi M, Schwartz PJ, Towbin JA, Vincent GM, Zhang L. Long-QT syndrome after age 40. Circulation. 2008 Apr 29;117(17):2192-201. doi: 10.1161/CIRCULATIONAHA.107.729368. Epub 2008 Apr 21. PMID 18427134
- [Background] Vaglio M, Couderc JP, McNitt S, Xia X, Moss AJ, Zareba W. A quantitative assessment of T-wave morphology in LQT1, LQT2, and healthy individuals based on Holter recording technology. Heart Rhythm. 2008 Jan;5(1):11-8. doi: 10.1016/j.hrthm.2007.08.026. Epub 2007 Aug 28. PMID 18180017
- [Background] Couderc JP, Vaglio M, Xia X, McNitt S, Wicker P, Sarapa N, Moss AJ, Zareba W. Impaired T-amplitude adaptation to heart rate characterizes I(Kr) inhibition in the congenital and acquired forms of the long QT syndrome. J Cardiovasc Electrophysiol. 2007 Dec;18(12):1299-305. doi: 10.1111/j.1540-8167.2007.00960.x. Epub 2007 Oct 4. PMID 17916157
- [Background] Crotti L, Spazzolini C, Schwartz PJ, Shimizu W, Denjoy I, Schulze-Bahr E, Zaklyazminskaya EV, Swan H, Ackerman MJ, Moss AJ, Wilde AA, Horie M, Brink PA, Insolia R, De Ferrari GM, Crimi G. The common long-QT syndrome mutation KCNQ1/A341V causes unusually severe clinical manifestations in patients with different ethnic backgrounds: toward a mutation-specific risk stratification. Circulation. 2007 Nov 20;116(21):2366-75. doi: 10.1161/CIRCULATIONAHA.107.726950. Epub 2007 Nov 5. PMID 17984373
- [Background] Moss AJ, Shimizu W, Wilde AA, Towbin JA, Zareba W, Robinson JL, Qi M, Vincent GM, Ackerman MJ, Kaufman ES, Hofman N, Seth R, Kamakura S, Miyamoto Y, Goldenberg I, Andrews ML, McNitt S. Clinical aspects of type-1 long-QT syndrome by location, coding type, and biophysical function of mutations involving the KCNQ1 gene. Circulation. 2007 May 15;115(19):2481-9. doi: 10.1161/CIRCULATIONAHA.106.665406. Epub 2007 Apr 30. PMID 17470695
- [Background] Daubert JP, Zareba W, Rosero SZ, Budzikowski A, Robinson JL, Moss AJ. Role of implantable cardioverter defibrillator therapy in patients with long QT syndrome. Am Heart J. 2007 Apr;153(4 Suppl):53-8. doi: 10.1016/j.ahj.2007.01.025. PMID 17394903
- [Background] Seth R, Moss AJ, McNitt S, Zareba W, Andrews ML, Qi M, Robinson JL, Goldenberg I, Ackerman MJ, Benhorin J, Kaufman ES, Locati EH, Napolitano C, Priori SG, Schwartz PJ, Towbin JA, Vincent GM, Zhang L. Long QT syndrome and pregnancy. J Am Coll Cardiol. 2007 Mar 13;49(10):1092-8. doi: 10.1016/j.jacc.2006.09.054. Epub 2007 Feb 27. PMID 17349890
- [Background] Treherne JM, Woodward SK, Varga ZM, Ritchie JM, Nicholls JG. Restoration of conduction and growth of axons through injured spinal cord of neonatal opossum in culture. Proc Natl Acad Sci U S A. 1992 Jan 1;89(1):431-4. doi: 10.1073/pnas.89.1.431. PMID 1729714
- [Background] Couderc JP, McNitt S, Xia J, Zareba W, Moss AJ. Repolarization morphology in adult LQT2 carriers with borderline prolonged QTc interval. Heart Rhythm. 2006 Dec;3(12):1460-6. doi: 10.1016/j.hrthm.2006.08.009. Epub 2006 Aug 10. PMID 17161789
- [Background] Tan HL, Bardai A, Shimizu W, Moss AJ, Schulze-Bahr E, Noda T, Wilde AA. Genotype-specific onset of arrhythmias in congenital long-QT syndrome: possible therapy implications. Circulation. 2006 Nov 14;114(20):2096-103. doi: 10.1161/CIRCULATIONAHA.106.642694. Epub 2006 Nov 6. PMID 17088455
- [Background] Goldenberg I, Moss AJ, Zareba W, McNitt S, Robinson JL, Qi M, Towbin JA, Ackerman MJ, Murphy L. Clinical course and risk stratification of patients affected with the Jervell and Lange-Nielsen syndrome. J Cardiovasc Electrophysiol. 2006 Nov;17(11):1161-8. doi: 10.1111/j.1540-8167.2006.00587.x. Epub 2006 Aug 14. PMID 16911578
- [Background] Zareba W. Genotype-specific ECG patterns in long QT syndrome. J Electrocardiol. 2006 Oct;39(4 Suppl):S101-6. doi: 10.1016/j.jelectrocard.2006.05.017. Epub 2006 Sep 11. PMID 16963070
- [Background] Hobbs JB, Peterson DR, Moss AJ, McNitt S, Zareba W, Goldenberg I, Qi M, Robinson JL, Sauer AJ, Ackerman MJ, Benhorin J, Kaufman ES, Locati EH, Napolitano C, Priori SG, Towbin JA, Vincent GM, Zhang L. Risk of aborted cardiac arrest or sudden cardiac death during adolescence in the long-QT syndrome. JAMA. 2006 Sep 13;296(10):1249-54. doi: 10.1001/jama.296.10.1249. PMID 16968849
- [Background] Goldenberg I, Mathew J, Moss AJ, McNitt S, Peterson DR, Zareba W, Benhorin J, Zhang L, Vincent GM, Andrews ML, Robinson JL, Morray B. Corrected QT variability in serial electrocardiograms in long QT syndrome: the importance of the maximum corrected QT for risk stratification. J Am Coll Cardiol. 2006 Sep 5;48(5):1047-52. doi: 10.1016/j.jacc.2006.06.033. Epub 2006 Jul 7. PMID 16949500
- [Background] Karp JM, Moss AJ. Dental treatment of patients with long QT syndrome. J Am Dent Assoc. 2006 May;137(5):630-7. doi: 10.14219/jada.archive.2006.0259. PMID 16739543
- [Background] Goldenberg I, Moss AJ, Maron BJ, Dick AW, Zareba W. Cost-effectiveness of implanted defibrillators in young people with inherited cardiac arrhythmias. Ann Noninvasive Electrocardiol. 2005 Oct;10(4 Suppl):67-83. doi: 10.1111/j.1542-474X.2005.00070.x. PMID 16274418
- [Background] Goldenberg I, Moss AJ, Zareba W. Sudden cardiac death without structural heart disease: update on the long QT and Brugada syndromes. Curr Cardiol Rep. 2005 Sep;7(5):349-56. doi: 10.1007/s11886-005-0088-1. PMID 16105490
- [Background] Zareba W, Moss AJ, Daubert JP, Hall WJ, Robinson JL, Andrews M. Implantable cardioverter defibrillator in high-risk long QT syndrome patients. J Cardiovasc Electrophysiol. 2003 Apr;14(4):337-41. doi: 10.1046/j.1540-8167.2003.02545.x. PMID 12741701
- [Background] Zareba W, Moss AJ. Long QT syndrome in children. J Electrocardiol. 2001;34 Suppl:167-71. doi: 10.1054/jelc.2001.28863. PMID 11781951
- [Background] Zhang L, Timothy KW, Vincent GM, Lehmann MH, Fox J, Giuli LC, Shen J, Splawski I, Priori SG, Compton SJ, Yanowitz F, Benhorin J, Moss AJ, Schwartz PJ, Robinson JL, Wang Q, Zareba W, Keating MT, Towbin JA, Napolitano C, Medina A. Spectrum of ST-T-wave patterns and repolarization parameters in congenital long-QT syndrome: ECG findings identify genotypes. Circulation. 2000 Dec 5;102(23):2849-55. doi: 10.1161/01.cir.102.23.2849. PMID 11104743
- [Background] Moss AJ. Long QT Syndromes. Curr Treat Options Cardiovasc Med. 2000 Aug;2(4):317-322. doi: 10.1007/s11936-996-0005-y. PMID 11096536
- [Background] Burattini L, Zareba W, Rashba EJ, Couderc JP, Konecki J, Moss AJ. ECG features of microvolt T-wave alternans in coronary artery disease and long QT syndrome patients. J Electrocardiol. 1998;31 Suppl:114-20. doi: 10.1016/s0022-0736(98)90302-8. PMID 9988014
- [Background] Zareba W, Moss AJ, Konecki J. TU wave area-derived measures of repolarization dispersion in the long QT syndrome. J Electrocardiol. 1998;30 Suppl:191-5. doi: 10.1016/s0022-0736(98)80074-5. PMID 9535499
- [Background] Zareba W, Moss AJ. Dispersion of repolarization. Relation to heart rate and repolarization duration. J Electrocardiol. 1995;28 Suppl:202-6. doi: 10.1016/s0022-0736(95)80057-3. PMID 8656112
- [Background] Moss AJ, Robinson JL. The long-QT syndrome Genetic considerations. Trends Cardiovasc Med. 1992 May-Jun;2(3):81-3. doi: 10.1016/1050-1738(92)90010-P. PMID 21239264
- [Background] Moss AJ, Robinson JL. Long QT syndrome. Heart Dis Stroke. 1992 Sep-Oct;1(5):309-14. No abstract available. PMID 1344123